CLINICAL TRIAL: NCT01616524
Title: A Phase 3, Randomized, Double-Blind, Controlled Study Evaluating the Efficacy and Safety of Peginterferon Lambda-1a, With and Without Daclatasvir, Compared to Peginterferon Alfa-2a, Each in Combination With Ribavirin, in the Treatment of Naïve Genotype 2 and 3 Chronic Hepatitis C Subjects
Brief Title: Safety and Efficacy Study of Pegylated Interferon Lambda With and Without Daclatasvir, Compared to Pegylated Interferon Alfa, Plus Ribavirin in Subjects With Hepatitis C Genotype 2 and 3
Acronym: PRINCIPAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI452-017; 2011-004885-14 (EudraCT Number)
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C Virus (HCV)
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon lambda-1a; peginterferon alfa-2a; Ribavirin; daclatasvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: pegIFNλ + Ribavirin + Placebo matching Daclatasvir (Experimental)
  Interventions: Biological: Pegylated interferon lambda (pegIFNλ); Drug: Ribavirin; Drug: Placebo matching Daclatasvir
- Arm 2: pegIFNλ + Ribavirin + Daclatasvir (Experimental)
  Interventions: Biological: Pegylated interferon lambda (pegIFNλ); Drug: Ribavirin; Drug: Daclatasvir
- Arm 3: pegIFNα-2a + Ribavirin + Placebo matching Daclatasvir (Experimental)
  Interventions: Biological: Pegylated interferon alfa-2a (pegIFNα-2a); Drug: Ribavirin; Drug: Placebo matching Daclatasvir

INTERVENTIONS:
Biological: Pegylated interferon lambda (pegIFNλ) — Syringe, Subcutaneous, 180 μg, Once weekly, 24 weeks
  Other Names: BMS-914143
  Arms: Arm 1: pegIFNλ + Ribavirin + Placebo matching Daclatasvir
Biological: Pegylated interferon lambda (pegIFNλ) — Syringe, Subcutaneous, 180 μg, Once weekly, 12 weeks
  Other Names: BMS-914143
  Arms: Arm 2: pegIFNλ + Ribavirin + Daclatasvir
Biological: Pegylated interferon alfa-2a (pegIFNα-2a) — Syringe, Subcutaneous, 180 μg, Once weekly, 24 weeks
  Other Names: Pegasys
  Arms: Arm 3: pegIFNα-2a + Ribavirin + Placebo matching Daclatasvir
Drug: Ribavirin — Tablets, Oral, 400 mg, Twice daily, 24 weeks
  Other Names: Ribasphere
  Arms: Arm 1: pegIFNλ + Ribavirin + Placebo matching Daclatasvir; Arm 3: pegIFNα-2a + Ribavirin + Placebo matching Daclatasvir
Drug: Ribavirin — Tablets, Oral, 400 mg, Twice daily, 12 weeks
  Other Names: Ribasphere
  Arms: Arm 2: pegIFNλ + Ribavirin + Daclatasvir
Drug: Daclatasvir — Tablets, Oral, 60 mg, Once daily, 12 weeks
  Other Names: BMS-790052
  Arms: Arm 2: pegIFNλ + Ribavirin + Daclatasvir
Drug: Placebo matching Daclatasvir — Tablets, Oral, 0 mg, Once daily, 12 weeks
  Arms: Arm 1: pegIFNλ + Ribavirin + Placebo matching Daclatasvir; Arm 3: pegIFNα-2a + Ribavirin + Placebo matching Daclatasvir

SUMMARY:
The purpose of this study is to determine if 24 weeks of treatment with Pegylated Interferon Lambda plus Ribavirin and 12 weeks of treatment with Pegylated Interferon Lambda plus Ribavirin and Daclatasvir will be safe and effective for treatment of hepatitis C compared to 24 weeks of treatment with Pegylated Interferon Alfa-2a plus Ribavirin

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Chronic hepatitis C, Genotype 2 or 3
* Naïve to prior anti-HCV therapy

Exclusion Criteria:

* Infected with HCV other than Genotype 2 or 3
* Positive Hepatitis B surface antigen (HBsAg), or Human immunodeficiency virus-1 (HIV-1)/HIV-2 antibody at screening
* Evidence of liver disease other than HCV
* Active substance abuse
* Evidence of decompensated cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve Sustained Virologic Response at post-treatment follow-up week 12 (SVR12) | Post-treatment follow-up week 12

SECONDARY OUTCOMES:
Proportion of subjects with Rapid virologic response (RVR) [undetectable Hepatitis C virus (HCV) Ribonucleic acid (RNA)] | On-treatment Week 4
Proportion of subjects with treatment emergent cytopenic abnormalities (anemia as defined by Hb < 10 g/dL, neutropenia as defined by ANC < 750 mm3 or thrombocytopenia as defined by platelets < 50,000 mm3) | Up to week 12 or week 24
  Hb = Hemoglobin ANC = Absolute neutrophil count
Proportion of subjects with on-treatment interferon-associated flu-like symptoms (as defined by pyrexia or chills or pain) | Up to week 12 or week 24
Proportion of subjects with on-treatment musculoskeletal symptoms (as defined by arthralgia or myalgia or back pain) | Up to week 12 or week 24
Proportion of subjects with Sustained Virologic Response at post-treatment follow-up week 24 (SVR24) by treatment group | Post-treatment week 24
Proportion of subjects with on-treatment Serious adverse events (SAEs) | Up to week 12 or week 24
Proportion of subjects with dose reductions | Up to week 12 or week 24
Proportion of subjects who discontinue due to Adverse events (AEs) | Up to week 12 or week 24
Proportion of subjects with SVR12 in subjects with genotype-3 (GT-3) chronic HCV infection | Post-treatment follow-up week 12
Proportion of subjects with on-treatment constitutional symptoms (fatigue or asthenia) | Up to week 12 or week 24

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (105):
- United States (18):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Precision Research Institute, Llc, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - University Of California, San Francisco/Sf General Hospital, San Francisco, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Orlando Immunology Center, Orlando, Florida
  - Orlando Infectious Disease Center, Orlando, Florida
  - Gastrointestinal Specialists Of Georgia, Marietta, Georgia
  - The Queen'S Liver Center, Honolulu, Hawaii
  - Henry Ford Hospital, Detroit, Michigan
  - Carolinas Medical Center, Charlotte, North Carolina
  - Consultants For Clinical Research, Cincinnati, Ohio
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - University Of Pittsburgh Medical Center, Ctr For Liver Diseases, Pittsburgh, Pennsylvania
  - Texas Clinical Research Institute, Llc, Arlington, Texas
  - St. Luke'S Episcopal Hospital - Baylor College Of Medicine, Houston, Texas
  - Clinical Research Centers Of America, Murray, Utah
- Argentina (7):
  - Local Institution, Autonoma, Buenos Aires
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, Quilmes, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Prov de Santa Fe, Santa Fe Province
- Australia (14):
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Concord, New South Wales
  - Local Institution, Darlinghurst, New South Wales
  - Local Institution, Randwick, New South Wales
  - Local Institution, Westmead Nsw, New South Wales
  - Local Institution, Brisbane, Queensland
  - Local Institution, Greenslopes, Queensland
  - Local Institution, Herston, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Clayton Vic, Victoria
  - Local Institution, Fitzroy, Victoria
  - Local Institution, Melbourne, Victoria
  - Local Institution, Parville, Victoria
  - Local Institution, Fremantle, Western Australia
- Belgium (3):
  - Local Institution, Brussels
  - Local Institution, Leuven
  - Local Institution, Liège
- Local Institution, Santiago, Santiago Metropolitan, Chile
- Local Institution, Hus, Finland
- France (4):
  - Local Institution, Clichy
  - Local Institution, Créteil
  - Local Institution, Montpellier
  - Local Institution, Nice
- Greece (2):
  - Local Institution, Athens
  - Local Institution, Thessaloniki
- Hong Kong (2):
  - Local Institution, Hong Kong
  - Local Institution, Tai Po
- Italy (4):
  - Local Institution, Florence
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Novara
- Japan (18):
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Kitakyushu, Fukuoka
  - Local Institution, Hiroshima, Hiroshima
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kobe, Hyōgo
  - Local Institution, Tsuchiura-shi, Ibaraki
  - Local Institution, Takamatsu, Kagawa-ken
  - Local Institution, Kagoshima, Kagoshima-ken
  - Local Institution, Kawasaki-shi, Kanagawa
  - Local Institution, Miyazaki, Miyazaki
  - Local Institution, Okayama, Okayama-ken
  - Local Institution, Saga, Saga-ken
  - Local Institution, Iruma-gun, Saitama
  - Local Institution, Saitama, Saitama
  - Local Institution, Bunkyo-ku, Tokyo
  - Local Institution, Minato-ku, Tokyo
  - Local Institution, Musashino-shi, Tokyo
  - Local Institution, Wakayama, Wakayama
- Mexico (6):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Distrito Federal, Mexico City
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Tlalpan, Mexico City
  - Local Institution, Guadalajara
  - Local Institution, Mexico City
- Netherlands (2):
  - Local Institution, Amsterdam
  - Local Institution, Leiden
- Local Institution, Auckland, New Zealand
- Russia (7):
  - Local Institution, Chelyabinsk
  - Local Institution, Irkutsk
  - Local Institution, Krasnoyarsk
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Samara
  - Local Institution, Smolensk
- Local Institution, Singapore, Singapore
- South Korea (6):
  - Local Institution, Busan
  - Local Institution, Daegu
  - Local Institution, Gyeonggi-do
  - Local Institution, Gyeongsangnam-do
  - Local Institution, Incheon
  - Local Institution, Seoul
- Taiwan (4):
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
  - Local Institution, Tainan
  - Local Institution, Yunlin
- United Kingdom (4):
  - Local Institution, Hull, Humberside
  - Local Institution, Nottingham, Nottinghamshire
  - Local Institution, Birmingham, West Midlands
  - Local Institution, London

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx